CLINICAL TRIAL: NCT04525768
Title: Characteristic of Patients With Gastroesophageal Varices and Portal Cavernoma
Brief Title: Gastroesophageal Varices in Cavernoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, XiaoquanHUANG, Resident, Shanghai Zhongshan Hospital
Other Study IDs: ZS-cavernoma-EGV
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Gastroesophageal Varices; Myeloproliferative Neoplasm; Portal Caver Cavernoma; Portal Hypertension
Keywords: portal hypertension; gastroesophageal varices; jak2 mutation; myeloproliferative Neoplasm; portal caver cavernoma
MeSH Terms: conditions — Myeloproliferative Disorders; Hypertension, Portal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JAK2 mutation Group: Patients with portal caver cavernoma and gastroesophageal varices and JAK2 Mutation.
  Interventions: Diagnostic Test: JAK2 mutation test
- Portal caver cavernoma Group: Patients with portal caver cavernoma and gastroesophageal varices without JAK2 Mutation.
  Interventions: Diagnostic Test: JAK2 mutation test

INTERVENTIONS:
Diagnostic Test: JAK2 mutation test — Patients with portal caver cavernoma will be divided into two groups by the result of JAK2 mutation test

SUMMARY:
Myeloproliferative neoplasms (MPNs), including polycythemia vera, essential thrombocythemia, and primary myelofibrosis, may lead to gastroesophageal varices. The quality of life, morbidity, and mortality of MPN patients mainly depend on disease-related symptoms, thromboembolic and hemorrhagic complications. Previous studies have shown that JAK2 V617F has a prominent role in vascular risk and MPN-associated gastroesophageal varices. Portal vein thrombosis and portal cavernoma frequently occur in the MPN population and the management of gastroesophageal varices in these patients are sometimes technically difficult. The aim of this study is to investigate the the characteristics of patients with gastroesophageal varices and portal caver cavernoma with or without JAK2 mutation.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients aged 18-75
* diagnosed as portal hypertension and portal cavernoma by contrast-enhanced computed tomography
* underwent JAK2 mutation test

Exclusion Criteria:

* combined known etiologies of chronic liver disease, including hepatitis, primary biliary cirrhosis, schistosomiasis, and non-alcoholic fatty liver disease.
* other factors judged by the investigator that may affect the safety of the subject or the compliance of the trial. Such as serious illnesses (including mental illness) that require combined treatment, serious laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed with portal cavernoma and gastric and/or esophageal varices and underwent JAK2 mutation test.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
History of variceal bleeding | 1 day (the same time as diagnosis)
  Have a history of the occurrence of gastroesophageal variceal bleeding

SECONDARY OUTCOMES:
1-year death rate | 1 year
  1-year death rate
Complications of portal hypertension | 1 year
  The concurrence of complications of portal hypertension (ascites, infections, variceal bleeding, et al)

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Reilly CR, Babushok DV, Martin K, Spivak JL, Streiff M, Bahirwani R, Mondschein J, Stein B, Moliterno A, Hexner EO. Multicenter analysis of the use of transjugular intrahepatic portosystemic shunt for management of MPN-associated portal hypertension. Am J Hematol. 2017 Sep;92(9):909-914. doi: 10.1002/ajh.24798. Epub 2017 Jul 26. PMID 28543980
- [Result] Yan M, Geyer H, Mesa R, Atallah E, Callum J, Bartoszko J, Yee K, Maganti M, Wong F, Gupta V. Clinical features of patients with Philadelphia-negative myeloproliferative neoplasms complicated by portal hypertension. Clin Lymphoma Myeloma Leuk. 2015 Jan;15(1):e1-5. doi: 10.1016/j.clml.2014.04.004. Epub 2014 Jun 11. PMID 25027569